CLINICAL TRIAL: NCT04043702
Title: Combination of Topiramate(Conviban) and Empagliflozin(Jardiance) is Considered a Good Option for the Treatment of Obesity
Brief Title: Combination of Topiramate and Empagliflozin is Considered a Good Option for the Treatment of Obesity
Status: Completed | Type: Observational
Sponsor: Ministry of Health and Population, Egypt (Other Government)
Responsible Party: Principal Investigator, mahmoud younis, Principal Investigator, Cairo University
Other Study IDs: 12345678
Record Dates: First submitted 2019-07-19; First posted 2019-08-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2019-08

CONDITIONS: Obesity
Keywords: obesity; drug combination; empagliflozin(jardiance); topiramate(conviban)
MeSH Terms: conditions — Obesity | interventions — empagliflozin; Topiramate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- on topiramate: "topiramate", "conviban®" group vs no treatment ( control group).
  Interventions: Drug: The intervention being studied
- on empagliflozine: "empagliflozine", "jardiance®" vs no treatment ( control group).
  Interventions: Drug: The intervention being studied
- on topiramate plus empagliflozine: all patients' vs no treatment ( control group).
  Interventions: Drug: The intervention being studied
- no treatment: all patients' vs no treatment ( control group).
  Interventions: Drug: The intervention being studied

INTERVENTIONS:
Drug: The intervention being studied — Intervention Other Names have not been specified
  Other Names: "empagliflozine", "jardiance®"); "topiramate", "conviban®"

SUMMARY:
The aim was to show if a combination of topiramate and empagliflozin have the greatest weight decreasing effect in comparison to each drug alone and to group with no treatment( control group).

.

DETAILED DESCRIPTION:
The aim was to show if a combination of topiramate and empagliflozin have the greatest weight decreasing effect in comparison to each drug alone and to group with no treatment( control group).

Materials and methods 200 obese patients 4 groups. had been monitored in a private clinic, each group 50 patients number, with 35 females and 15 males who were already on treatment.

ELIGIBILITY:
Inclusion Criteria:

1. stable weight in the previous 6 months.
2. a sedentary lifestyle.
3. no history of diabetes mellitus.
4. taking medication that affects appetite, or weight within the past 6 months

Exclusion Criteria:

1. severe anemia
2. hypothyroidism and hyperthyroidism
3. Diabetes mellitus
4. moderate to severe liver or kidney disease
5. body mass index less than 30

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: obese peoples , age from 35 to 55 years
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2019-07-20 (Actual); Study Completion 2019-07-29 (Actual)

PRIMARY OUTCOMES:
change in weight | 6 months
  weight measurement

CONTACTS AND LOCATIONS:
Overall Officials: mahmoud younis, M.S, Principal Investigator — egyptian ministry of health
Locations (1):
- Mahmoud Younis, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No